CLINICAL TRIAL: NCT03414073
Title: Comparative Evaluation of the Plaque Removal Efficacy and Patient Acceptability of the Knotted Floss Technique With Conventional Flossing Technique and Interdental Brushing in Type II Gingival Embrasures - A Clinical Crossover Study
Brief Title: Evaluation of Plaque Removal Efficacy & Patient Acceptability of Knotted Floss Technique in Type II Gingival Embrasures
Acronym: KF-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uttaranchal Dental & Medical Research Institute (Other)
Responsible Party: Principal Investigator, Aaron Gomes, Prof & Head, Dept of Periodontics & Oral Implantology, Uttaranchal Dental & Medical Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UttaranchalDMRI_KF-II
Record Dates: First submitted 2018-01-20; First posted 2018-01-29 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Oral Hygiene; Dental Devices, Home Care
Keywords: dental floss; gingival embrasure; oral hygiene; interdental brush

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allotted to three groups. each group will undergo three treatment phases with an in-between washout phase.In each treatment phase the group subjects will test a different intervention
Who Masked: Outcomes Assessor
Masking Description: Only the Principal investigator will know the intervention being done by subject. The outcome investigator(assessor) will be unaware (blinded) to which intervention the subject is undertaken
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group A Phase 1 (Sham Comparator): Conventional flossing technique using commercially available Reach® Floss One third of sample are randomly assigned to Group A and are to utilise conventional finger flossing technique in the first phase of 4-weeks. For the conventional flossing technique the subjects will wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "C" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure.
  Interventions: Device: Conventional flossing technique
- Group B Phase 1 (Active Comparator): Knotted floss technique using an improvised flossing technique by putting a knot in commercially available Reach® Floss One third of sample are randomly assigned to Group B and are to utilise knotted floss technique in the first phase of 4-weeks, twice daily. The subjects will use the supplied floss lengths having a simple knot in the middle and will perform the same way as the conventional finger flossing technique, except that the insertion of floss will have to be in the non-knotted area and during the to and fro movements the knotted area of the floss will have to be engaged in the interdental area.
  Interventions: Device: Knotted floss technique
- Group C Phase 1 (Sham Comparator): Conventional interdental brushing technique using Thermoseal® Proxa ns interdental brushes One third of sample are randomly assigned to Group C and are to utilise conventional interdental brushing technique in the first phase of 4-weeks twice daily. The subjects will gently insert the brush into the interdental area with an inclination akin to the angle of the interdental gums (gingiva), and perform to and fro buccal to lingual movements and a little apico-coronal movement such that the gingiva is not impinged, and finally removing the brush out buccally.
  Interventions: Device: Conventional Interdental Brushing
- Group A Phase 2 (Active Comparator): Knotted floss technique using an improvised flossing technique by putting a knot in commercially available Reach® Floss After a washout period of 2 weeks, those from Group A will use the knotted floss technique in the second phase for a period of 4 weeks, twice daily. The subjects will use the supplied floss lengths having a simple knot in the middle and will perform the same way as the conventional finger flossing technique, except that the insertion of floss will have to be in the non-knotted area and during the to and fro movements the knotted area of the floss will have to be engaged in the interdental area.
  Interventions: Device: Knotted floss technique
- Group B Phase 2 (Sham Comparator): Conventional interdental brushing technique using Thermoseal® Proxa ns interdental brushes After a washout period of 2 weeks, those from Group B will use the conventional interdental brushing technique in the second phase for a period of 4 weeks, twice daily. The subjects will gently insert the brush into the interdental area with an inclination akin to the angle of the interdental gums (gingiva), and perform to and fro buccal to lingual movements and a little apico-coronal movement such that the gingiva is not impinged, and finally removing the brush out buccally.
  Interventions: Device: Conventional Interdental Brushing
- Group C Phase 2 (Sham Comparator): Conventional flossing technique using commercially available Reach® Floss After a washout period of 2 weeks, those from Group C will use the conventional finger flossing technique in the second phase for a period of 4 weeks, twice daily. For the conventional flossing technique the subjects will wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "C" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure.
  Interventions: Device: Conventional flossing technique
- Group A Phase 3 (Sham Comparator): Conventional interdental brushing technique using Thermoseal® Proxa ns interdental brushes After a washout period of 2 weeks, those from Group A will use the conventional interdental brushing technique in the third phase for a period of 4 weeks, twice daily. The subjects will gently insert the brush into the interdental area with an inclination akin to the angle of the interdental gums (gingiva), and perform to and fro buccal to lingual movements and a little apico-coronal movement such that the gingiva is not impinged, and finally removing the brush out buccally.
  Interventions: Device: Conventional Interdental Brushing
- Group B Phase 3 (Sham Comparator): Conventional flossing technique using commercially available Reach® Floss After a washout period of 2 weeks, those from Group B will use the conventional finger flossing technique in the third phase for a period of 4 weeks, twice daily. For the conventional flossing technique the subjects will wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "C" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure.
  Interventions: Device: Conventional flossing technique
- Group C Phase 3 (Active Comparator): Knotted floss technique using an improvised flossing technique by putting a knot in commercially available Reach® Floss After a washout period of 2 weeks, those from Group C will use the knotted floss technique in the third phase for a period of 4 weeks, twice daily. The subjects will use the supplied floss lengths having a simple knot in the middle and will perform the same way as the conventional finger flossing technique, except that the insertion of floss will have to be in the non-knotted area and during the to and fro movements the knotted area of the floss will have to be engaged in the interdental area.
  Interventions: Device: Knotted floss technique

INTERVENTIONS:
Device: Knotted floss technique — The subjects use the knotted floss technique. In this modification of conventional flossing technique, a knot is tied in the floss at any distance in the middle third of the floss length. The floss is inserted past the interdental contact point by the conventional finger flossing technique in the non-knotted area and then during the 'to and fro movement' on the tooth surface cervical to contact point, the knotted area is engaged through the embrasure (Gomes et al 2016)
  Arms: Group A Phase 2; Group B Phase 1; Group C Phase 3
Device: Conventional flossing technique — The subject will wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "C" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure.
  Other Names: Finger Flossing; Conventional finger flossing technique
  Arms: Group A Phase 1; Group B Phase 3; Group C Phase 2
Device: Conventional Interdental Brushing — The subject will gently insert the interdental brush into the interdental area with an inclination akin to the angle of the interdental gums (gingiva), and perform to and fro buccal to lingual movements and a little apico-coronal movement such that the gingiva is not impinged, and finally removing the brush out buccally.
  Other Names: Interdental Brushes for interproximal cleaning
  Arms: Group A Phase 3; Group B Phase 2; Group C Phase 1

SUMMARY:
Removal and prevention of formation of dental plaque biofilms is the cornerstone of current hygiene regimens to prevent, reduce or even reverse the gingival and periodontal disease condition. In such endeavors of mechanical plaque removal, tooth-brushing and use of dental floss play an important role. Gomes et al have presented a modification in the use of knotted floss in wider embrasure areas. The modification in the dental floss has been done so as to increase the effective width of the floss. The purpose of this study is to compare the reduction of the clinical signs of plaque accumulation, gingival inflammation, gingival bleeding and gingival trauma in the area the knotted floss technique has been utilized versus the area where conventional flossing or interdental brush has been utilized in Type II gingival embrasures. Patients' acceptability of the knotted flossing technique will also be evaluated.

DETAILED DESCRIPTION:
Substantial evidence exists that show that effective plaque control leads to reduction in prevalence and severity of gingival inflammation. Use of toothbrush with dentifrice is a common mean for removing plaque on many tooth surfaces, research has shown that it cannot completely clean the interdental surfaces when used without other interproximal aids. Dental flossing is useful in cleaning interproximal surfaces of teeth from the contact point to the sulcus especially in Type I interdental embrasures. Interdental brushes are used by patients with sufficient space between their teeth or the Type II interdental embrasures. To make the dental floss effective in wide embrasure areas Gomes et al, have recently presented a modification in the technique of flossing and called it the 'Knotted Floss Technique'. Unpublished data by the same authors in a crossover study shows that knotted floss technique is equally safe and effective method for reducing plaque, inflammation and bleeding when compared to conventional finger flossing in Type I gingival embrasures.

The purpose of this study is to compare the reduction of the clinical signs of plaque accumulation, gingival inflammation and gingival trauma in type II gingival embrasures that the knotted floss technique has been used with similar embrasures that a conventional flossing technique has been used, as well as with identical type embrasures wherein an inter-dental brush has been utilized. Patients' acceptability of the knotted flossing technique will also be evaluated.

Materials and Methods:

Criteria for Sample Selection: For this triple phase, examiner blind, crossover clinical trial, a sample size of thirty individuals who were eighteen years and above will be randomly selected from the outpatients of the Department of Periodontology and Oral Implantology at the college hospital. The inclusion and exclusion criteria will be as described later. The trial will be conducted as per the guidelines in the WHO-Handbook for Good Clinical Practice and the research protocol is approved by the Institutional Ethics Committee of the college.

Design of Study: A sample size of thirty subjects will be selected based on the criteria above. Prior to commencement of the actual study, each volunteer will receive written and verbal instructions on the two techniques. Investigator 1 & 3 will demonstrate to the volunteers all 3-techniques on models, for ½hour counseling session, for 3 consecutive days. Each counseling session will have not more than 10 participants. The techniques demonstrated on models will be conventional finger flossing, knotted floss technique and cleaning of interdental area with interdental brush. The conventional finger flossing technique will be demonstrated to the volunteers as follows: to wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "C" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure. For the knotted floss technique, the volunteers will perform the same way as the conventional finger flossing technique, except that the insertion of floss will have to be in the non-knotted area and during the to and fro movements the knotted area of the floss will have to be engaged in the interdental area. When using the interdental brush, the volunteers will be demonstrated to gently insert the brush into the interdental area with an inclination akin to the angle of the interdental gums (gingiva), and perform to and fro buccal to lingual movements and a little apico-coronal movement such that the gingiva is not impinged, and finally removing the brush out buccally. On the 4th day, after both investigators will be separately satisfied with the volunteer's proficiency on models, with respect to each of the three techniques demonstrated, an informed consent will be taken and the volunteer will be enrolled as a subject into the 16-week, 3-phase crossover, single (examiner) blind study protocol with washout phases of 2-weeks each in-between the intervention phases. Failure by the volunteer to perform the techniques as instructed will mean another counseling session of 1-hour, followed by another check of proficiency by volunteer on models by the above investigators on subsequent day. If the investigators are not satisfied with the ability of the volunteer to perform any one of the 3 demonstrated techniques of interdental cleansing even after an extra counselling session, then the volunteer will not be recruited into the study protocol.

Investigator#1 will be randomly placed into three groups (Group A, Group B, Group C) by the draw of lots. Each group will participate in three treatment phases of 4-weeks each with a 2-week washout phase in between the 3-treatment phases. Group A will perform conventional finger flossing in 1st phase, followed by knotted floss technique and interdental brushing in the 2nd and 3rd treatment phase respectively. Group B will perform knotted floss technique, interdental brushing and conventional finger flossing in the 1st, 2nd and 3rd treatment phase respectively; while Group C will perform interdental brushing, conventional finger flossing and knotted floss technique in their 1st, 2nd, 3rd treatment phases respectively. Only the 1st investigator will be responsible for this allocation and coding of subjects to respective treatment groups and the other investigators will be blind as to which technique the subject will be assigned to. Each treatment phase will consist of 4-weeks of daily use of the assigned interdental cleansing technique. At the baseline appointment for each treatment phase, every subject will be given their assigned interdental cleansing products by the 1st investigator (only). Subjects assigned to conventional flossing will receive 60-pieces of waxed floss [Reach¬®-Johnson & Johnson Consumer Inc.], 15-centimeters in length each piece, equally divided in 3-bags [Ziplock®-S.C. Johnson & Son, Inc.]. Subjects assigned to knotted flossing aid will receive the same except that every floss thread will have a simple knot at around the middle. Subjects assigned to the interdental brush cleansing regimen will receive 60-pieces of interdental brushes [Thermoseal® Proxa ns interdental brushes-ICPA Health Products Ltd] equally divided in 3-bags, instead of the pieces of floss. Each subject will also receive a sample of toothbrush [Oral-B® Allrounder Soft Toothbrush-Procter & Gamble India Ltd.] and dentifrice [Colgate® Strong Teeth Dentifrice-Colgate-Palmolive Company Ltd.]. The subjects will be instructed to brush their teeth twice a day in their customary manner using the above toothbrush and dentifrice and will be cautioned not to use any other oral hygiene aid except for the assigned interdental cleansing device twice a day. The subjects will have to return to the 1st author any unused interdental cleansing product(s) at the end of the treatment phase. The 1st and 2nd treatment phase will be followed by a 'washout period'. During the washout period the subjects will be instructed to perform normal oral hygiene practices of tooth-brushing with dentifrice and refrain from using any floss, interdental brush or any additional plaque control aids. The "washout" period is designed so as to give subjects time to return to their original oral status and establish parity in baseline clinical measurements prior to starting the next treatment phase. Such a 'washout' in crossover-study design will allowed use of 50% lesser subjects.

Clinical evaluations: Clinical evaluations of all subjects will be done at 2-weekly intervals, namely baseline, 2-weeks and 4-weeks of each treatment phase. Both adjacent teeth and gingiva at test sites will be scored for the Rustogi Modification of Navy Plaque Index, Lobene's Modified Gingival Index, and Barnett's Modified Papillary Bleeding Index. The sequencing of examination is specifically chosen as plaque index, gingival index and bleeding index, so as to avoid the possibility that the plaque will be removed during the recording of the other two indices. A plaque disclosing agent will be used to identify the location and amount of plaque. Additionally, gingival trauma will also be assessed as presence or absence of signs of trauma in the marginal and papillary gingiva of adjacent teeth as per the methodology proposed by Carter-Hanson et al. The facial and lingual surfaces will be examined visually for gingival lacerations. Presence of laceration, floss cut, or demarcation line/indentation at the site will be scored as one, while a score of zero (0) will be recorded when there is absence of any signs of trauma. The score per subject will be obtained by totaling all scores and dividing by number of sites examined.

The indices will be recorded by investigators #2 & 4. Intra- and inter-examiner reliability will be recorded prior to commencement of the study and at 2-weekly intervals throughout the study. A rate of concordance will also be established. The study schedule will so be distributed, such that not more than six subjects reported for examination on any given day of the week. These two investigators will be blinded as to which technique the subject is using and the amount of unused floss if any at end of respective treatment phase.

Subject compliance: A compliance diary will also be given to each subject at the baseline appointment of each treatment phase and will be collected at the end of each phase by the investigator #1. The subjects will be instructed to record each interdental cleansing experience in this diary and any other event he/she will feel is significant. A patient satisfaction questionnaire will be answered by every subject at the end of the third and final treatment phase. Compliance or non-compliance by the subject will thus tried to be established by calculating the amount of any unused portion of interdental cleansing product and by the entries in the diary. Investigator #3 will contact the subjects after completion of the study to verify any unusual entries in the compliance diary or to ascertain the reasons of excess unused floss returned to the department if any.

Analysis of Data: Data will be recorded by investigator #2 &4 into coded case sheets per subject. This data after decoding by investigator #1 will be tabulated wherein the scores at respective time periods of conventional flossing technique from all three treatment groups, will be tabulated together and similarly those of knotted floss technique and interdental brushing. The scores for plaque, gingival inflammation, gingival bleeding and gingival trauma will be tabulated separately. The mean differences and standard deviations will be calculated. The mean differences of scores at respective time intervals of each of the index scored will be compared between the three interdental cleansing techniques by using the analysis of variance (ANOVA) and the paired sample test. This will determine the statistical difference between scores of the three different techniques whilst calculating a specific index at respective time interval. Also, a statistical analysis by paired t-test will be done of difference of scores recorded between 2-weeks and baseline, 4-weeks and baseline, 4-weeks and 2-weeks of that specific index within the same treatment technique. This will determine the improvement/worsening/no effect of respective scores of plaque, gingival inflammation, gingival bleeding and gingival trauma over a 4 week period while using the same interdental cleansing technique. The responses given by the patient to the end-study questionnaire will be aggregated and analyzed on a percentage scale to compare preference between each technique.

ELIGIBILITY:
Inclusion Criteria:

* have one Type II gingival embrasure in the premolar first molar area.
* full mouth Plaque Index score ≥1.8 (Silness and Loe 1964)
* full mouth Gingival Index ≥ 1.0 (Loe and Silness 1963)
* good general health,
* have all teeth present in quadrant being tested and opposing quadrant
* be available for a 16 week study period,
* be ready to abide with the study criteria,
* minimum education of grade 12

Exclusion Criteria:

* have used in previous 2-months oral hygiene aids other than tooth-brushing like dental flossing, mouthwashes and water jet irrigating systems
* habit of unilateral mastication for ≥2 months,
* medical history of diabetes mellitus, hepatitis, pregnancy or requiring any antibiotic prophylaxis,
* having drug history in preceding two months of use of antibiotics, hormonal supplements, steroids, non steroidal anti-inflammatory medications, oral contraceptives or any drug that influence gingival tissue,
* taking part in any other clinical or drug trial including taking part in other study groups related to the evaluation of knotted floss technique,
* having physical handicap limiting the ability for oral hygiene and effective use of dental floss,
* had orthodontic treatment
* having gross dental caries
* having advanced periodontitis (more than one pocket ≥ 6mm),
* had active periodontal treatment like scaling, root planing, curettage, periodontal surgery in the previous 8-weeks,
* had any adverse oral habit like smoking, tobacco chewing or habits of self gingival mutilation,
* had history of trauma or surgery to the jaws.
* teeth adjacent to the embrasure area selected are having proximal caries or gross occlusal caries, or having proximal restorations, crowns, onlays or inlays.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Rustogi modification of Navy Plaque Index - 4-weeks | 4 weeks
  Rustogi modification of Navy Plaque Index will be assessed at 4-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Lobene's Modified Gingival Index - 4-weeks | 4 weeks
  Lobene's Modified Gingival Index will be assessed at 4-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Barnett's Modified Papillary Bleeding Index - 4 Weeks | 4 weeks
  Barnett's Modified Papillary Bleeding Index will be assessed at 4-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Gingival Trauma Index (as Described by Carter-Hanson et al 1996) - 4-weeks | 4 weeks
  Gingival Trauma Index (as Described by Carter-Hanson et al 1996) will be assessed at 4-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3

SECONDARY OUTCOMES:
Rustogi modification of Navy Plaque Index - Baseline | Baseline
  Rustogi modification of Navy Plaque Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Lobene's Modified Gingival Index - baseline | baseline
  Lobene's Modified Gingival Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Barnett's Modified Papillary Bleeding Index - baseline | baseline
  Barnett's Modified Papillary Bleeding Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Gingival Trauma Index (as Described by Carter-Hanson et al 1996) - baseline | baseline
  Gingival Trauma Index (as Described by Carter-Hanson et al 1996) will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Rustogi Modification of Navy Plaque Index - 2 Weeks | 2 weeks
  Rustogi modification of Navy Plaque Index will be assessed at 2-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Lobene's Modified Gingival Index - 2-weeks | 2 weeks
  Lobene's Modified Gingival Index will be assessed at 2-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Barnett's Modified Papillary Bleeding Index - 2 Weeks | 2 weeks
  Barnett's Modified Papillary Bleeding Index will be assessed at 2-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3
Gingival Trauma Index (as Described by Carter-Hanson et al 1996) - 2-weeks | 2 weeks
  Gingival Trauma Index (as Described by Carter-Hanson et al 1996) will be assessed at 2-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group C Phase 1, Group A Phase 2, Group B Phase 2, Group C Phase 2, Group A Phase 3, Group B Phase 3 and Group C Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Aaron F Gomes, MDS, Principal Investigator — Uttaranchal Dental & Medical Research Institute, Dehradun, India
Locations (1):
- Dept of Periodontics & Oral Implantology; Uttaranchal Dental and Medical Reserach Institute, Dehradun, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hansen F, Gjermo P. The plaque-removing effect of four toothbrushing methods. Scand J Dent Res. 1971;79(7):502-6. No abstract available. PMID 5289846
- [Background] Loe H, Schiott CR, Karring G, Karring T. Two years oral use of chlorhexidine in man. I. General design and clinical effects. J Periodontal Res. 1976 Jun;11(3):135-44. doi: 10.1111/j.1600-0765.1976.tb00061.x. No abstract available. PMID 133217
- [Background] Loe H. Mechanical and chemical control of dental plaque. J Clin Periodontol. 1979 Dec;6(7):32-6. doi: 10.1111/j.1600-051x.1979.tb02116.x. No abstract available. PMID 295293
- [Background] Anerud A, Loe H, Boysen H, Smith M. The natural history of periodontal disease in man. Changes in gingival health and oral hygiene before 40 years of age. J Periodontal Res. 1979 Nov;14(6):526-40. doi: 10.1111/j.1600-0765.1979.tb00255.x. No abstract available. PMID 161591
- [Background] Choo A, Delac DM, Messer LB. Oral hygiene measures and promotion: review and considerations. Aust Dent J. 2001 Sep;46(3):166-73. doi: 10.1111/j.1834-7819.2001.tb00277.x. PMID 11695154
- [Background] Claydon NC. Current concepts in toothbrushing and interdental cleaning. Periodontol 2000. 2008;48:10-22. doi: 10.1111/j.1600-0757.2008.00273.x. No abstract available. PMID 18715352
- [Background] Carter-Hanson C, Gadbury-Amyot C, Killoy W. Comparison of the plaque removal efficacy of a new flossing aid (Quik Floss) to finger flossing. J Clin Periodontol. 1996 Sep;23(9):873-8. doi: 10.1111/j.1600-051x.1996.tb00626.x. PMID 8891940
- [Background] Asadoorian J. Flossing: Canadian Dental Hygienists Association position statement. Canadian J Dent Hygiene 2006;40(3):1-10.
- [Background] Christou V, Timmerman MF, Van der Velden U, Van der Weijden FA. Comparison of different approaches of interdental oral hygiene: interdental brushes versus dental floss. J Periodontol. 1998 Jul;69(7):759-64. doi: 10.1902/jop.1998.69.7.759. PMID 9706852
- [Background] Gjermo P, Flotra L. The effect of different methods of interdental cleaning. J Periodontal Res. 1970;5(3):230-6. doi: 10.1111/j.1600-0765.1970.tb00722.x. No abstract available. PMID 4254187
- [Background] Bellamy P, Barlow A, Puri G, Wright KI, Mussett A, Zhou X. A new in vivo interdental sampling method comparing a daily flossing regime versus a manual brush control. J Clin Dent. 2004;15(3):59-65. PMID 15688960
- [Background] Shibly O, Ciancio SG, Shostad S, Mather M, Boardman TJ. Clinical evaluation of an automatic flossing device vs. manual flossing. J Clin Dent. 2001;12(3):63-6. PMID 11505962
- [Background] Schmid M. Plaque control. In: Carranza F, editor. Glickman's clinical periodontology. 6th ed. Philadelphia: W.B Saunders Company; 1984:689-690.
- [Background] Carr MP, Rice GL, Horton JE. Evaluation of floss types for interproximal plaque removal. Am J Dent. 2000 Aug;13(4):212-4. PMID 11763934
- [Background] Van de Weijden GA, Slot DE. Interdental oral hygiene: the evidence. In: Bartold PM, Jin LJ, eds. Multi-Disciplinary Management of Periodontal Disease. Adelaide, South Australia: Asian Pacific Society of Periodontology; 2012:16-33. Available at: http://www.apsperio.org/APSPProceedings2011.pdf. Accessed January 15, 2018.
- [Background] Gomes AF, Meru S, Rekhi A. Knotted floss technique. J Advanced Res Dent Oral Health 2016;1(1):6-7.
- [Background] Gomes AF, Rekhi A, Meru S, Chahal G. Evaluation of plaque removal efficacy and patient acceptability of knotted floss technique in type I gingival embrasures. U.S. National Library of Medicine. ClinicalTrials.gov identifier: NCT02931994. Available at: https://clinicaltrials.gov/ct2/show/NCT02931994.htm.
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Adwazi K, Crawley F, Idänpään-Heikkilä JE, et al. World Health Organization. Handbook for good clinical research practice (GCP): guidance for implementation. WHO Library Cataloguing-in-Publication Data. France. 2005. Available at http://apps.who.int/medicinedocs/pdf/whozip13e/whozip13e.pdf. Accessed April 6, 2015.
- [Background] Rustogi KN, Curtis JP, Volpe AR, Kemp JH, McCool JJ, Korn LR. Refinement of the Modified Navy Plaque Index to increase plaque scoring efficiency in gumline and interproximal tooth areas. J Clin Dent. 1992;3(Suppl C):C9-12. PMID 1306676
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Barnett M, Ciancio S, Mather M. The modified papillary bleeding index: comparison with gingival index during the resolution of gingivitis. J Prev Dent 1980; 6:135-138.
- [Background] Gomes AF, S M, Rekhi A. Letter to the Editor: Re: Reducing Dental Plaque and Gingivitis With 0.6% Cortex Ilicis Rotundae Toothpaste: A Randomized, Double-Masked Clinical Trial. J Periodontol. 2017 Jan;88(1):1. doi: 10.1902/jop.2016.160513. Epub 2016 Nov 4. No abstract available. PMID 27809632